CLINICAL TRIAL: NCT01879852
Title: Muscle Weakness and Post-traumatic Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00060374; K01HD052713 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Meniscectomy
Keywords: Quadriceps strength; Knee; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Rehabilitation (Active Comparator): Standard meniscectomy rehabilitation including knee range of motion and strengthening exercises.
  Interventions: Behavioral: Standard rehabilitation
- Standard Rehabilitation + Quadriceps intensive strengthening (Experimental): The intervention includes high-intensity neuromuscular electrical stimulation and eccentric exercises for the quadriceps muscle in addition to the standard rehabilitation protocol.
  Interventions: Behavioral: Quadriceps intensive strengthening; Behavioral: Standard rehabilitation

INTERVENTIONS:
Behavioral: Quadriceps intensive strengthening — Quadriceps intensive strengthening includes high-intensity neuromuscular electrical stimulation to the quadriceps muscle for 10 minutes and overload to the the eccentric phase of quadriceps strengthening exercises.
  Arms: Standard Rehabilitation + Quadriceps intensive strengthening
Behavioral: Standard rehabilitation — Standard rehabilitation will include interventions for typical knee impairments (effusion, knee motion deficits, lower extremity muscle weakness, and gait deviations) as well as advanced rehabilitation interventions as indicated (jump and agility exercises)

SUMMARY:
This is a single-center, randomized, single-blind (evaluator) study. Enrolled patients had a traumatic meniscal tear and underwent meniscectomy. The study included 6 weeks (12 visits) of standard or quadriceps intensive rehabilitation. The objective of the study was to determine the effect of quadriceps intensive rehabilitation on knee function and articular cartilage.

ELIGIBILITY:
Inclusion Criteria:

1. traumatic onset meniscal tear (i.e. specific mechanism of injury)
2. meniscectomy surgery performed within 12 months of index injury
3. meniscal tear confirmed at the time of surgery
4. subject anticipates living in close proximity to Gainesville for one year following surgery.

Exclusion Criteria:

1. bilateral injury
2. concomitant ligamentous injury
3. previous knee injury
4. articular cartilage defect > Grade II on Outerbridge scale
5. patellofemoral joint pain > 3/10 with activity
6. lower limb alignment > 5 degrees of valgus or varus
7. contraindication to an MR examination including: a pacemaker, metal implants which are not MR compatible, pregnancy and severe claustrophobia.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terese Chmielewski, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 subjects were consented to the study. During pre-surgery (baseline) testing, 2 subjects were found not to have a meniscal tear (inclusion criterion) and were withdrawn from the study. Total number of subjects meeting eligibility criteria was 27.
Period: Overall Study
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening
Started | 14 | 13
Completed | 12 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The target number of participants was determined statistically from preliminary data on primary outcome measures. The final population was based on feasibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (5.2) | 18.3 (2.8) | 20.4 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 176.9 (8.5) | 180.1 (8.8) | 178.5 (8.7)
Weight [Mean (Standard Deviation); unit: kg] | 78.7 (13.2) | 100.9 (30.1) | 89.8 (26.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in International Knee Documentation Committee (IKDC) Subjective Knee Form Score
Description: The IKDC is a measure of self-reported knee function and includes items related to symptoms and functional activity. Responses on the IKDC subjective knee form will be recorded on hard-copy and the summary score computed. The highest (best) possible score is 100 points and the lowest (worst) possible score is 0 points.
Time Frame: Baseline (pre-surgery) to 7 weeks post-surgery (post-intervention)
Population: 2 subjects in the Standard Rehabilitation group did not complete the intervention or post-treatment testing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening
Number analyzed (Participants) | 12 | 13
units on a scale | 22.2 (21.6) | 20.6 (21.1)

2. Primary Outcome: Change in Tibial Articular Cartilage Volume
Description: A magnetic resonance image (MRI) of the knee will be acquired and software will be used to quantify tibial articular cartilage volume.
Time Frame: Baseline (pre-surgery) to 1 year post-surgery
Population: 2 subjects in the Standard Rehabilitation group did not complete the intervention or post-treatment testing. Images were not analyzable for one subject in the Standard+Quadriceps Intensive Strengthening group.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening
Number analyzed (Participants) | 12 | 11
percentage change from baseline | 0.18 (3.21) | -1.24 (4.27)

3. Secondary Outcome: Single Leg Forward Hop Index
Description: Three trials of the single leg forward hop will be collected on each side. Distance will be averaged across trials. The single leg hop index will be computed as [(distance on the surgical side/distance on the non-surgical side) *100]
Time Frame: 7 weeks post-surgery (post-intervention)
Population: 2 subjects in the Standard Rehabilitation group did not complete the intervention or post-treatment testing. 2 subjects in the Standard Rehabilitation group and 1 subject in the Standard + Quadriceps Intensive Strengthening group did not complete hop testing.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening
Number analyzed (Participants) | 10 | 12
percentage | 87.1 (15.2) | 90.1 (10.9)

4. Secondary Outcome: Change in Urinary Concentrations of C-terminal Crosslinking Telopeptide of Type II Collagen (CTX-II)
Description: CTX-II is a biomarker of Type II collagen degradation. Early-morning, second void, fasting urine samples will be collected and stored. Concentrations of CTX-II will be determined with enzyme-linked immunosorbent assay, corrected for creatine concentration, and log-transformed. Creatinine concentration will also be determined with enzyme-linked immunosorbent assay.
Time Frame: Baseline (pre-surgery) to 7 weeks post-surgery (post-intervention)
Population: 2 subjects in the Standard Rehabilitation group did not complete the intervention or post-treatment testing.
Measure: Mean (Standard Deviation); unit: log (ng/mmol)
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening
Number analyzed (Participants) | 12 | 13
log (ng/mmol) | 0.01 (0.18) | -0.11 (0.13)

ADVERSE EVENTS:
Arm/Group | Standard Rehabilitation | Standard Rehabilitation + Quadriceps Intensive Strengthening
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

LIMITATIONS AND CAVEATS:
Difficulty with subject recruitment due to concomitant injury with meniscal tear

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No